CLINICAL TRIAL: NCT01228994
Title: Testing the GABAergic Hypothesis of Nicotine Dependence: a Randomized Clinical Trial of Baclofen
Brief Title: Baclofen for Smoking Cessation in a Non-Psychiatric Population
Acronym: Baclofen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because of difficulties recruiting subjects.
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Tobacco Control Research Initiative (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Prinicipal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1632009
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Nicotine Dependence
Keywords: smoking cessation treatment; baclofen; Smoking cessation counselling
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baclofen 30 mg/day (Active Comparator): Baclofen medication
  Interventions: Drug: Baclofen 30 mg/day
- Placebo pill (Placebo Comparator): placebo pill
  Interventions: Drug: placebo pill
- Baclofen 60 mg/day (Active Comparator): Baclofen medication high dose
  Interventions: Drug: Baclofen 60 mg/day

INTERVENTIONS:
Drug: Baclofen 30 mg/day — Baclofen 30 mg/day for 8 weeks with 2 week induction and 2 week decrease
  Other Names: Lioresal, Kemstro
  Arms: Baclofen 30 mg/day
Drug: placebo pill — placebo pill
  Arms: Placebo pill
Drug: Baclofen 60 mg/day — baclofen 60 mg/day for 8 weeks with 2 week induction and 2 week decrease
  Other Names: Lioresal, Kemstro
  Arms: Baclofen 60 mg/day

SUMMARY:
The primary hypothesis for this study is that, in nicotine-dependent tobacco smokers, baclofen will be superior to placebo for smoking abstinence measures.

The secondary hypothesis is that subjects assigned to the baclofen groups will exhibit higher rates of medication compliance (i.e. take the medication as directed for the trial period) than those in the placebo group.

The tertiary hypothesis is that baclofen will lead to significant reductions in tobacco withdrawal and craving ratings as compared to placebo.

DETAILED DESCRIPTION:
This study will test a new medication strategy designed to help smokers quit. It will evaluate Baclofen, a drug currently approved and available in Canada as a myorelaxant. Forty five nicotine-dependent smokers will enroll in this study. Fifteen will receive placebo (inactive pill), fifteen will receive baclofen 30 mg/day, and fifteen will receive baclofen 60 mg/day. Once enrolled, subjects will visit CAMH on a weekly basis for assessment of smoking behaviour, a brief health check (vitals, BP and AE screening), delivery of brief individual smoking cessation counselling, and collection of breath, blood and urine samples (as scheduled) to a) measure levels of nicotine and its metabolites, b) conduct pregnancy and tox testing. The medication phase of this study lasts 12 weeks. Two follow-up visits will be scheduled at week 13 and at six months after trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (18 years or older).
* Meet DSM-IV criteria for nicotine dependence,
* Smoke ≥10 cigarettes/day,
* Baseline FTND score ≥4, CO level ≥10,
* have had at least one failed quit attempt in the past and are motivated to quit within 30 days of initial intake.
* No previous use of medication for smoking cessation in 1 month prior to randomization.
* BMI between 15 and 40 inclusive.

Exclusion Criteria:

* Meet DSM-IV criteria for a current diagnosis of major depressive disorder, panic disorder or post-traumatic stress disorder, or a current or past history of bipolar disorder or schizophrenia
* Have a past history of major depression, with historical evidence of suicidal or homicidal behaviour, or psychotic symptom,
* Have abused alcohol or other drugs of abuse (cocaine, opiates, benzodiazepines, etc) in 3 months prior to randomization
* Demonstrate serious medical conditions, unstable cardiovascular disease, significant blood abnormalities)
* Are pregnant, are trying to become pregnant or are currently breastfeeding
* Baclofen hypersensitivity .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence for 7 days at end of treatment | end of treatment week 10
  At end of treatment subjects will report smoking consumption for past 7 days. Subject are considered abstinent based on self report and verfied by CO level (<10 PPM)
Abstinent rate: last four weeks of trial | last 4 weeks of trial (week 7 to 10)
  subjects report cigarette consumption during the last 4 weeks of the clinical trial.
  abstinence rates are verifed by CO < 10 PPM
abstinence rate: for past 7 days at 6 month followup | 6 month followup
  Subject are asked to attend a 6 month followup. At this time subjects will be asked to report their cigarette consumption for the past 7 days.
  abstinence is based on this self report and verified by CO levels <10 PPM

SECONDARY OUTCOMES:
Tiffany Questionnaire of Smoking Urges | screen, week 1,4,7,10, abd 6 month followup
  tobacco craving is monitored at different time points of the trial
Minnesota Nicotine Withdrawal Scale | Screen, week 1,4,7,10 and 6 month followup
  This scale assesses symptoms of tobacco withdrawal including nicotine craving, irritability, anziety, difficulty conentrating, restlessness, headaches, fatigue, increased appetite, weight gain, and insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health- 33 Russell St, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research